CLINICAL TRIAL: NCT07312604
Title: Evaluating the Therapeutic Efficacy of Intra-lesional Immunotherapy Against Recalcitrant Tinea Cruris & Corporis: a Pilot Study
Brief Title: A Pilot Study to Evaluate the Therapeutic Efficacy of Intra-Lesional Immunotherapy in Patients Aged 10-60 Years With Recalcitrant Tinea Cruris and Corporis
Acronym: IL-ImmuneRTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abeer Mohamed Abdelaziz Elkholy (Other)
Collaborators: Mansoura University Hospital (Other)
Responsible Party: Sponsor-Investigator, Abeer Mohamed Abdelaziz Elkholy, Professor of Dermatology, Faculty of Medicine, Mansoura University, Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.25.11.3446
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Tinea Corporis; Tinea Cruris
Keywords: Tinea Cruris; Tinea Corporis; Recalcitrant Dermatophytosis; Intra-Lesional Immunotherapy; Pilot Clinical Study; Dermatophyte Treatment
MeSH Terms: conditions — Tinea; Tinea Cruris | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-Lesional Immunotherapy (Experimental): All participants with recalcitrant tinea cruris and/or tinea corporis will receive intra-lesional immunotherapy. There is no comparator or placebo group. Male and female participants are included in the same arm and will be analyzed as subgroups.Intra-Lesional Immunotherapy
  Interventions: Biological: Intra-Lesional MMR Immunotherapy

INTERVENTIONS:
Biological: Intra-Lesional MMR Immunotherapy — Participants will receive intra-lesional immunotherapy using the measles-mumps-rubella (MMR) vaccine. The vaccine will be injected into the active borders of affected lesions every 2 weeks for a total duration of 6 weeks. Clinical assessment of lesion extent and symptoms, particularly pruritus, will be performed at baseline and at each visit. If partial clinical improvement is observed after the initial 6 weeks but complete resolution is not achieved, the treatment course may be extended for an additional 6 weeks, with a maximum of six intra-lesional injection sessions.
  Other Names: MMR Vaccine; Measles-Mumps-Rubella Vaccine; Priorix®

SUMMARY:
This pilot study will test intra-lesional immunotherapy (MMR vaccine) injections as a treatment for recalcitrant tinea cruris and corporis in patients aged 10-60 years who have not improved with standard antifungal treatments.

*Eligibility: Participants must have recalcitrant tinea, defined as:

* Rapid progression or large areas of skin affected,
* Infection in multiple family members, especially females and children
* Rapid relapse after prior treatment
* Suspected resistant T. indotineae (based on travel history or contact with affected individuals from high-prevalence regions)
* Failure of at least 2 courses of systemic antifungal therapy in the past 3 months

Treatment: Patients will receive intra-lesional MMR vaccine injections into the active borders of affected lesions every 2 weeks for up to 6 weeks. If partial improvement occurs but complete clearance is not achieved, the course may be repeated for another 6 weeks. Pulse itraconazole will be given during the first 2 weeks.

Monitoring: At each study visit, clinicians will assess the extent of affected skin and monitor symptoms particularly itching. Safety will be closely observed, including injection-site reactions, fever, initial flare of lesions, and any rare serious allergic reactions.

Goal: To evaluate the safety and effectiveness of intra-lesional MMR immunotherapy for patients with tinea that has been difficult to treat.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 - 60 years.
* Evidence of recalcitrant tinea e.g. (rapid progression & large areas affected of the body, affection of more than one family members especially females & children, rapid relapse after treatment, suspicion of resistant T. indotineae strain by history of traveling abroad & contact with Indians or contact with a case coming from travel & with contact to Indians.
* Patients failed at least 2 courses of systemic antifungal therapy in the last 3 months.
* Safe contraception during the study (for females in the childbearing period).

Exclusion Criteria:

* Pregnant or lactating women, as well as women of childbearing potential not using an effective method of contraception.
* Age <10 years or > 60 years.
* Immunocompromised patients e.g. (uncontrolled DM or HIV patients).
* Naïve patients without previous systemic antifungal treatment.
* Unreliable patients.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in affected body surface area (BSA) from baseline | Assessed at each study visit (every 2 weeks) up to 6 weeks, with extension up to 12 weeks if improvement is notice after initial 6 weeks, but complete resolution isn't achieved.
  The primary efficacy endpoint is the percent reduction in the total body surface area affected by recalcitrant tinea (cruris and/or corporis), assessed by clinical examination at each study visit. This measure evaluates the improvement in lesion extent and treatment response over time.

SECONDARY OUTCOMES:
Safety and Tolerability: Incidence and severity of treatment-emergent adverse events | Monitored continuously throughout the initial 6-week treatment period, with continued observation up to 12 weeks if a second course is administered.
  All adverse events (AEs) occurring during the study including injection site reactions, fever or initial flare, increased pruritus as well as severe reactions (anaphylaxis or angioedema) will be systematically monitored and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt